CLINICAL TRIAL: NCT03738150
Title: A Phase 2a Single-Arm, Open-Label, Multicenter Exploratory Study to Assess the Effects of Sotatercept (ACE-011) for the Treatment of Pulmonary Arterial Hypertension
Brief Title: A Study of Sotatercept for the Treatment of Pulmonary Arterial Hypertension
Acronym: SPECTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A011-10; 7962-002 (Other: Merck)
Record Dates: First submitted 2018-11-02; First posted 2018-11-13 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotatercept (Experimental): Each participant will receive SOC plus sotatercept at a dose of 0.3 mg/kg SC for Cycle 1. (Each cycle will be 21 days.) From Cycle 2 through Cycle 9, the dose will be escalated to 0.7 mg/kg SC. Dosing will be every three weeks during the 24-week treatment period and 18-month extension period.
  Interventions: Biological: Sotatercept; Other: SOC

INTERVENTIONS:
Biological: Sotatercept — Sotatercept injection
  Other Names: ACE-011
Other: SOC — SOC therapy refers to combination therapy consisting of drugs from two or more of the following drug classes: an endothelin-receptor antagonist (ERA), a phosphodiesterase 5 (PDE5) inhibitor, a soluble guanylate cyclase stimulator, and/or a prostacyclin analogue or receptor agonist.

SUMMARY:
This study evaluates the effect of sotatercept (ACE-011) in adults with pulmonary arterial hypertension (PAH). Each eligible participant will receive standard of care (SOC) plus sotatercept (ACE-011) for a 24-week treatment period, followed by an 18-month extension period, and an 8-week follow-up period.

DETAILED DESCRIPTION:
This is a Phase 2a, single-arm, open-label, multicenter exploratory study to determine the effects of sotatercept plus SOC in adults with WHO functional class III PAH.

All eligible participants will receive SOC plus sotatercept at a starting dose level of 0.3 mg/kg by subcutaneous (SC) injection for Cycle 1 and escalating to 0.7 mg/kg at Cycle 2 for the remainder of the treatment period. Participants will be required to attend clinic visits once every three weeks for the 24-week treatment period and once every three weeks for the 18-month extension period to perform one or more protocol specified evaluations. Evaluations include hemodynamic measures collected during right heart catheterization (RHC) with invasive cardiopulmonary exercise test (iCPET), and cardiac magnetic resonance imaging (MR), 6-minute walk distance (6MWD), pharmacokinetic parameters, pharmacodynamic parameters, anti-drug antibody testing, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Documented findings on RHC at any time prior to Screening consistent with a diagnosis of World Health Organization (WHO) pulmonary hypertension Group 1: PAH of any of the following subtypes:

   * Idiopathic PAH
   * Heritable PAH
   * Drug- or toxin-induced PAH
   * PAH associated with connective tissue disease
   * PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following shunt repair
3. Symptomatic pulmonary hypertension classified as WHO functional class III
4. Screening RHC documenting a minimum PVR of ≥ 4 Wood units
5. Pulmonary function tests within 6 months prior to Screening as follows:

   1. Total lung capacity > 70% predicted; or if between 60% to 70% predicted, or not possible to be determined, confirmatory high-resolution computed tomography (CT) indicating no more than mild interstitial lung disease per investigator interpretation or
   2. Forced expiratory volume (first second) (FEV1)/forced vital capacity (FVC) > 70% predicted
   3. For subjects with a history of lobectomy or pneumonectomy, and for whom there are no population-based normalization methods, assessment based on residual lung volume will be permitted to assess eligibility.
6. Ventilation-perfusion (VQ) scan (or, if unavailable, a negative CT pulmonary angiogram [CTPA] or pulmonary angiography result), any time prior to Screening or conducted during Screening Period with normal or low probability result
7. 6MWD ≥ 100 and ≤ 550 meters repeated twice during Screening Period and both values within 15% of each other, calculated from the highest value
8. Combination PAH therapy at stable (per investigator) dose levels for at least 90 days prior to Cycle 1 Day 1 (C1D1)

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Started or stopped receiving any general supportive therapy for pulmonary hypertension (e.g., diuretics, oxygen, anticoagulants, digoxin) within 60 days prior to C1D1 (Cycle 1 Day 1)
2. Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to C1D1
3. History of atrial septostomy within 180 days prior to Screening
4. History of more than mild obstructive sleep apnea that is untreated
5. History of portal hypertension or chronic liver disease, defined as mild to severe hepatic impairment (Child-Pugh Classes A to C)
6. History of human immunodeficiency virus infection-associated PAH
7. Prior exposure to sotatercept (ACE-011) or luspatercept (ACE-536)
8. Uncontrolled systemic hypertension as evidenced by sitting systolic BP > 160 mm Hg or sitting diastolic BP > 100 mm Hg during Screening after a period of rest
9. Systolic BP < 90 mm Hg during Screening or at baseline
10. History of known pericardial constriction
11. Electrocardiogram (ECG) with QTcF > 480 msec during Screening or C1D1
12. History of personal or family history of long QTc syndrome or sudden cardiac death
13. History of restrictive or constrictive cardiomyopathy
14. Left ventricular ejection fraction < 45% on echocardiogram performed within 6 months of Screening OR pulmonary capillary wedge pressure (PCWP) > 15 mm Hg on RHC during baseline evaluation
15. Any current symptomatic coronary disease (myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain in the past 6 months prior to Screening)
16. Acutely decompensated heart failure within 30 days prior to C1D1, as per investigator assessment
17. Significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC; Jonathan Lu, MD, Study Director — Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA
Locations (4):
- United States (4):
  - The University of Arizona, Tucson, Arizona
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Waxman AB, Systrom DM, Manimaran S, de Oliveira Pena J, Lu J, Rischard FP. SPECTRA Phase 2b Study: Impact of Sotatercept on Exercise Tolerance and Right Ventricular Function in Pulmonary Arterial Hypertension. Circ Heart Fail. 2024 May;17(5):e011227. doi: 10.1161/CIRCHEARTFAILURE.123.011227. Epub 2024 Apr 4. PMID 38572639

RESULTS

PARTICIPANT FLOW:
Groups:
- Sotatercept: Each participant received standard of care (SOC) plus sotatercept at a dose of 0.3 mg/kg by subcutaneous (SC) injection during Cycle 1. (Each cycle was 21 days.) From Cycle 2 through Cycle 9, the dose was escalated to 0.7 mg/kg SC. Dosing occurred once every 3 weeks during the 24-week treatment period and 18-month extension period.
Period: Base Study
Arm/Group | Sotatercept
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Extension Study
Arm/Group | Sotatercept
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sotatercept
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (15.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Peak Oxygen Uptake (VO2 max) at Baseline [Mean (Standard Deviation); unit: mL/min/kg] — Each participant's VO2 max was measured by an invasive cardiopulmonary exercise test (iCPET) at baseline. Population: All participants who completed treatment period, had iCPET assessment and cardiac magnetic resonance imaging (MRI) at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at End Of Treatment (EOT), with no major protocol deviations.
  mL/min/kg
    number analyzed (Participants) | 17
    (all) | 11.02 (3.204)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Oxygen Uptake (VO2 Max) at 24 Weeks
Description: Each participant's VO2 max was measured by an invasive cardiopulmonary exercise test (iCPET) at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at End Of Treatment (EOT), with no major protocol deviations.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
mL/min/kg | 1.28 (2.628)

2. Secondary Outcome: Change From Baseline in Right Ventricular Stroke Volume (RV SV) at 24 Weeks
Description: Each participant's RV SV was measured by cardiac MRI at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
mL | -27.306 (26.5786)

3. Secondary Outcome: Change From Baseline in Right Ventricular End-Systolic Volume (RV ESV) at 24 Weeks
Description: Each participant's RV ESV was measured by cardiac MR imaging at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
mL | -39.151 (22.5544)

4. Secondary Outcome: Change From Baseline in Right Ventricular End-Diastolic Volume (RV EDV) at 24 Weeks
Description: Each participant's RV EDV was measured by cardiac MR imaging at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
mL | -66.459 (37.3311)

5. Secondary Outcome: Percent Change From Baseline in Right Ventricular Ejection Fraction (RV EF) at 24 Weeks
Description: Each participant's RV EF was measured by cardiac MR imaging at baseline and at 24 weeks.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
Percent change | -1.3 (8.48)

6. Secondary Outcome: Change From Baseline in Right Ventricular Stroke Volume Index (RV SVI) at 24 Weeks
Description: Each participant's RV SVI was measured by cardiac MR imaging at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
mL/m^2 | -15.073 (14.8219)

7. Secondary Outcome: Change From Baseline in Right Ventricular (RV) Mass at 24 Weeks
Description: Each participant's RV mass was measured by cardiac MR imaging at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
grams | -6.240 (13.3558)

8. Secondary Outcome: Change From Baseline in Ventilatory Efficiency (VE/VCO2 Slope) at 24 Weeks
Description: VE/VCO2 slope refers to the slope of the regression line of Minute Ventilation (VE) in liters/minute in the Y-axis and corresponding carbon dioxide production per minute (VCO2) in liters/minute in the X-axis plotted with multiple measurements taken during exercise. Each participant's VE/VCO2 slope at peak exercise was measured by an iCPET at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
Unitless | -8.87 (12.298)

9. Secondary Outcome: Change From Baseline in Cardiac Index at 24 Weeks
Description: Each participant's cardiac index at peak exercise was measured by iCPET at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and who had data for Change from Baseline in Cardiac Index at 24 Weeks.
Measure: Mean (Standard Deviation); unit: Liter/min/m^2
Arm/Group | Sotatercept
Number analyzed (Participants) | 16
Liter/min/m^2 | 0.411 (1.1944)

10. Secondary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure at 24 Weeks
Description: Each participant's pulmonary arterial pressure at peak exercise was measured by iCPET at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and who had data for Change from Baseline in Mean Pulmonary Arterial Pressure at 24 Weeks.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sotatercept
Number analyzed (Participants) | 16
mmHg | -14.9 (13.22)

11. Secondary Outcome: Change From Baseline in Arteriovenous O2 Content Difference (Ca-vO2) at 24 Weeks
Description: Each participant's Ca-vO2 at peak exercise was measured by iCPET at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and who had data for Change from Baseline in Ca-vO2 at 24 Weeks.
Measure: Mean (Standard Deviation); unit: mL/100 mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
mL/100 mL | 0.63 (2.131)

12. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at 24 Weeks
Description: Each participant's PVR, at resting supine, was measured by right heart catheterization (RHC) at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and who had data for Change from Baseline in PVR at 24 Weeks.
Measure: Mean (Standard Deviation); unit: dynes*sec/cm^5
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
dynes*sec/cm^5 | -305.728 (313.9827)

13. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at 24 Weeks
Description: 6MWD is measured by an exercise test known as 6MWT that assesses aerobic capacity and endurance. It measures the distance covered over a time of 6 minutes and is used as an outcome measure by which to compare changes in performance capacity. Each participant's 6MWD was measured at baseline and at 24 weeks. An increase in the distance walked during the 6MWT indicates improvement in basic mobility.
Time Frame: Baseline and 24 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and who had data for Change from Baseline in 6MWD at 24 Weeks.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sotatercept
Number analyzed (Participants) | 16
meters | 66.35 (85.659)

14. Secondary Outcome: Change From Baseline in Concentration of Amino-Terminal Brain Natriuretic Propeptide (NT-proBNP) at 24 Weeks
Description: Each participant's laboratory biomarkers N-terminal prohormone brain-type natriuretic peptide (NT-proBNP) or brain-type natriuretic peptide (BNP) were measured at baseline and at 24 weeks.
Time Frame: Baseline and 24 Weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and had data for Change from Baseline in Concentration of NT-proBNP at 24 Weeks.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
pg/mL | -623.1 (840.56)

15. Secondary Outcome: Change From Baseline in WHO (World Health Organization) Functional Class at 24 Weeks
Description: The World Health Organization (WHO) functional class describes how severe a person's pulmonary hypertension symptoms are. There are four different classes - I is the mildest and IV the most severe form of pulmonary hypertension.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: WHO functional class
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
WHO functional class | -0.76 (0.903)

16. Secondary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 24 weeks
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept
Number analyzed (Participants) | 21
Participants | 20

17. Secondary Outcome: Number of Participants Who Experienced One or More Events Indicative of Clinical Worsening of Pulmonary Arterial Hypertension (PAH)
Description: Events that indicate clinical worsening of PAH include death, need for and/or worsening-related listing for lung and/or heart transplant, need to initiate an approved PAH SOC rescue therapy, PAH-specific hospitalization, or functional deterioration (worsened WHO Functional Class AND 15% decrease in 6MWD).
Time Frame: Up to 102 weeks
Population: All participants who completed treatment period, had iCPET assessment and cardiac MRI at 24 weeks or ended treatment early and had iCPET assessment and cardiac MRI at EOT, with no major protocol deviations; and who had data for Number of Participants Who Experienced One or More Events Indicative of Clinical Worsening of PAH.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept
Number analyzed (Participants) | 17
Participants | 1

18. Secondary Outcome: Observed Trough Concentration (Ctrough) of Sotatercept at Cycle 9
Description: Ctrough is the plasma concentration of a drug prior to administration.
Time Frame: Day 1 of Cycle 9 (Each cycle was 21 days.)
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for Observed Ctrough of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 14
ng/mL | 5884.79 (2933.77)

19. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Sotatercept at Cycle 9
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The Cmax parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment and had at least 1 blood sample analyzed for PK, had data for Cmax of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
ng/mL | 9732.785 (2852.373)

20. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Sotatercept at Cycle 9
Description: Cmin is a measure of the minimum amount of drug in the plasma after the dose is given. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The Cmin parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for Cmin of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
ng/mL | 6234.303 (2466.046)

21. Secondary Outcome: Average Concentration (Cavg) of Sotatercept at Cycle 9
Description: Cavg is calculated by area under the plasma concentration versus dosing interval time curve at steady-state divided by the dosing interval. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The Cavg parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for Cavg of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
ng/mL | 8221.907 (2749.846)

22. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to T (AUC0-T) of Sotatercept at Cycle 9
Description: AUC0-T (area under the plasma concentration versus time curve from time zero after a dose is given to a period of one 21-day cycle) is a measure of the mean concentration levels of a drug in the plasma at steady state. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The AUC0-T parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for AUC0-T of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
ng*day/mL | 172659.953 (57746.622)

23. Secondary Outcome: Apparent Terminal Half-life (t1/2 ) of Sotatercept at Cycle 9
Description: t1/2 is the elimination half-life of study drug: the time it takes for half of the study drug in the blood plasma to dissipate. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The t1/2 parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for Apparent t1/2 of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
Days | 21.919 (5.861)

24. Secondary Outcome: Apparent Serum Clearance (CL) of Sotatercept at Cycle 9
Description: Apparent serum CL is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The apparent serum CL parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for Apparent Serum CL of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
Liters/day | 0.213 (0.077)

25. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Sotatercept at Cycle 9
Description: Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The Vz/F parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, and had data for Apparent Vz/F of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sotatercept
Number analyzed (Participants) | 15
Liters | 3.969 (1.078)

26. Secondary Outcome: Absorption Rate Constant (Ka) of Sotatercept at Cycle 9
Description: Ka is the proportionality constant that relates the rate of drug absorbed into the body. Ka is a value used to describe the rate at which a drug enters into the system. It is expressed in units of time. PopPK modeling approach was used to build a population PK model that captures the totality of the observed data from Cycles 1 to 9. The Ka parameter is derived from this preliminary popPK modeling.
Time Frame: Day 1 of each 21-day cycle: Cycles 1-9
Population: All participants who received at least 1 dose of study treatment, had at least 1 blood sample analyzed for PK, had data for Ka of Sotatercept at Cycle 9, and followed the dosing regimen.
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | Sotatercept
Number analyzed (Participants) | 14
1/day | 0.280 (0.035)

ADVERSE EVENTS:
Time Frame: Treatment period: Up to 24 weeks; Extension period: Up to 18 months plus 8-week follow-up period.
Description: The safety analysis population included all participants who received at least one dose of study treatment. The analysis population for All-Cause Mortality included all allocated participants.
Groups:
- Sotatercept Treatment Period: Each participant received standard of care (SOC) plus sotatercept at a dose of 0.3 mg/kg SC during Cycle 1. (Each cycle was 21 days.) For the remainder of the 24-week treatment period (Cycle 2 through Cycle 9), participants received an escalated dose of 0.7 mg/kg SC. Dosing occurred once every 3 weeks.
- Sotatercept Extension Period: Each participant received standard of care (SOC) plus sotatercept at a dose of 0.7 mg/kg SC once every 3 weeks during the 18-month extension period.
Arm/Group | Sotatercept Treatment Period | Sotatercept Extension Period
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/21 | 2/20
Other Adverse Events (participants affected / at risk) | 14/21 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept Treatment Period (N=21) | Sotatercept Extension Period (N=20)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept Treatment Period (N=21) | Sotatercept Extension Period (N=20)
Polycythaemia (Blood and lymphatic system disorders) | 3 (9) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 4 (4)
Complication associated with device (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (4) | 2 (2)
Pain (General disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7)
Dizziness (Nervous system disorders) | 2 (2) | 2 (4)
Headache (Nervous system disorders) | 3 (4) | 3 (3)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03738150/Prot_SAP_000.pdf